CLINICAL TRIAL: NCT05053334
Title: A Randomized Phase I, Double-Blinded, Parallel Comparative Assessment of PK, PD, Safety, and Immunogenicity of BP11 Versus US-Licensed Xolair® and EU Approved-Xolair® Following a Single 150 mg Dose SC Administration in Healthy Male Volunteers
Brief Title: Biosimilar Study Comparing PK, PD, Safety and Immunogencity of BP11 With US Licensed Xolair and EU Approved Xolair
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: CuraTeQ Biologics Private Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BP11-101
Record Dates: First submitted 2021-08-22; First posted 2021-09-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- BP11 (Proposed biosimilar) (Experimental): Subcutaneous injection of Omalizumab developed by CuraTeQ.
  Interventions: Drug: Omalizumab Prefilled Syringe
- US-Xolair (Active Comparator): Subcutaneous injection of Omalizumab licensed for use in USA
  Interventions: Drug: Omalizumab Prefilled Syringe
- EU-Xolair (Active Comparator): Subcutaneous injection of Omalizumab approved for use in Europe.
  Interventions: Drug: Omalizumab Prefilled Syringe

INTERVENTIONS:
Drug: Omalizumab Prefilled Syringe — 150mg/ml of Omalizumab prefilled syringe

SUMMARY:
A single dose, double blind comparative trial to assess the pharmacokinetics, pharmacodynamics, safety and immunogenicity of 3 different products (BP11, US-Xolair and EU-Xolair) containing 150mg of Omalizumab as subcutaneous injection in healthy male volunteers.

DETAILED DESCRIPTION:
The study will be conducted at 2 sites in New Zealand and 1 site in Australia.

A total of 165 healthy male subjects (55 subjects per arm) who meet the required entry criteria will be randomly assigned to one of 3 treatment groups in a 1:1:1 ratio to receive a single SC injection of either BP11, EU-Xolair, or US-Xolair.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent prior to any study-specific procedures, ability to understand, and willingness to comply with the study procedures, restrictions, and requirements as judged and confirmed by the Investigator.
2. Healthy adult male subjects, 18 to 55 years (both inclusive) of age at the time of signing informed consent.
3. Subjects who are considered healthy as determined by clinically acceptable findings of hematology, clinical chemistry, coagulation profile, urinalysis, and 12-lead ECG as per investigator's discretion.
4. Subject must agree to use a highly effective contraception as detailed in Appendix 1(Section 13.1) during the study period (starting from screening visit) and until 9 months after administration of BP11, Xolair® -EU or Xolair® -US by agreeing to use (with their female partner if she is of childbearing potential) 2 acceptable forms of contraception.
5. Subjects must refrain from donating sperm or fathering a child during the study period (starting from screening visit) and until 9 months after administration of BP11, Xolair®-EU or Xolair®-US administration by agreeing to use (with their female partner if she is of childbearing potential) 2 acceptable forms of contraception.

Exclusion Criteria:

1. Known history of hypersensitivity or allergic reactions to omalizumab or any of its excipients.
2. History of cardiovascular, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological, psychiatric or any other disease which in the opinion of the Investigator would make the subject inappropriate for study participation.
3. Abnormal and clinically relevant (in the opinion of the Investigator) vital signs, ECG, history of angina, exertional dyspnea, orthopnea, congestive heart failure, or myocardial infarction.
4. Major surgery or major trauma within past one year of screening or anticipated need for any surgery during the study duration.
5. Difficulty in blood sampling or difficulty in accessibility of veins.
6. History of significant alcohol abuse within 1 years prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
7. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
8. Subjects with positive drug test at screening or admission.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 165 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
To evaluate pharmacokinetic (PK) similarity of BP11 with US-Xolair and EU-Xolair and between US-Xolair and EU-Xolair | Upto 127 Days
  AUC0-inf will be evaluated
To evaluate PK similarity of BP11 with US-Xolair and EU-Xolair and between US-Xolair and EU-Xolair | Upto 127 Days
  Cmax will be evaluated

SECONDARY OUTCOMES:
To assess and compare non-primary PK parameters of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  AUC0-t
To assess and compare non-primary PK parameters of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Vd
To assess and compare non-primary PK parameters of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Tmax, T½
To assess and compare pharmacodynamics (PD) of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Free IgE levels will be assessed
To assess and compare pharmacodynamics (PD) of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Total IgE levels will be assessed
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Assessment of Vital signs-Blood pressure
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Assessment of Vital signs-Pulse rate
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Assessment of Vital signs-Body temperature
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Upto 127 Days
  Assessment of Vital signs-Respiratory rate
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Screening, Pre-dose (within 1 hour of drug administration) and post dose on day 3)
  Normal 12 Lead ECG (Ventricular rate)
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Screening, Pre-dose (within 1 hour of drug administration) and post dose on day 3)
  Normal 12 Lead ECG (PR interval)
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Screening, Pre-dose (within 1 hour of drug administration) and post dose on day 3)
  Normal 12 Lead ECG (QRS complex)
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Screening, Pre-dose (within 1 hour of drug administration) and post dose on day 3)
  Normal 12 Lead ECG (QT interval and QT interval corrected for heart rate using Bazett's formula)
Safety & tolerability of BP11 with US-Xolair and EU-Xolair | Pre-dose(0hour or within 1 hour prior of drug administration), post dose at 6hours, 12 hours and 24hours.
  Assessment of injection site reaction

CONTACTS AND LOCATIONS:
Locations (3):
- Q-Pharm Pty Ltd, Herston, Queens Land, Australia
- New Zealand (2):
  - Auckland Clinical Studies Ltd (NZCR OpCo Limited), Grafton, Auckland
  - Christchurch Clinical Studies Trust Ltd (NZCR OpCo Limited), Christchurch

IPD SHARING:
Plan to Share IPD: No